CLINICAL TRIAL: NCT00045357
Title: Phase I Study to Evaluate the Safety of Cellular Adoptive Immunotherapy Using Autologous CD4+ Antigen-Specific T Cell Clones for Patients With Metastatic Melanoma
Brief Title: Biological Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1585.00; FHCRC-1585.00; NCI-H02-0093; CDR0000256867 (Registry Identifier: PDQ)
Record Dates: First submitted 2002-09-06; First posted 2003-07-08 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop tumor cells from growing. Treating a person's white blood cells in the laboratory and reinfusing them may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of biological therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of autologous CD4+ antigen-specific T-cells for cellular adoptive immunotherapy in patients with metastatic melanoma.
* Determine the safety and toxicity of this regimen in these patients.
* Determine the duration of in vivo persistence of adoptively transferred CD4+ antigen-specific T-cell clones in these patients.

Secondary

* Determine the antitumor effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients undergo leukapheresis to collect peripheral blood mononuclear cells. CD4+ antigen-specific T-cell clones are generated over the next 2-3 months using immunogenic peptides MART1, tyrosinase, or gp100.

Patients receive autologous CD4+ antigen-specific T-cells IV over 30 minutes.

Cohorts of 3-6 patients receive escalating doses of autologous CD4+ antigen-specific T-cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed on days 1 and 3 post T-cell infusion, and then once weekly for 12 weeks.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma
* HLA type expressing one of the following class II alleles:

  * DRB1*0401
  * DRB1*0404
  * DRB1*1501
  * DPB1*0401
  * DPB1*0402
* Tumor expresses tyrosinase
* Tumor expressing NY-ESO-1 and are HLA type DP4, DP2, or DR7 allowed
* No CNS metastases

  * Prior CNS involvement allowed provided there is no evidence of CNS disease at least 2 months after treatment

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* Karnofsky 70-100%

Life expectancy

* More than 16 weeks

Hematopoietic

* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 30%

Hepatic

* SGOT no greater than 3 times upper limit of normal
* INR no greater than 1.5 due to hepatic dysfunction
* No significant hepatic dysfunction, defined as hepatic toxicity grade 2 or greater

Renal

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min
* Calcium no greater than 12 mg/dL

Cardiovascular

* No significant cardiac abnormalities*, defined by any 1 of the following:

  * Congestive heart failure
  * Clinically significant hypotension
  * Symptoms of coronary artery disease
  * Cardiac arrhythmias present on EKG requiring drug therapy NOTE: *Patients with a history of cardiovascular disease or any of the above abnormalities undergo a cardiac evaluation, including a cardiac stress test and/or echocardiogram

Pulmonary

* No clinically significant pulmonary dysfunction
* FEV1 at least 1.0 L OR
* FEV1 at least 60%
* DLCO at least 55% (corrected for hemoglobin)

Immunologic

* No acquired or hereditary immunodeficiency
* No autoimmune disease
* No active infection
* No oral temperature greater than 38.2 degrees C within the past 72 hours
* No systemic infection requiring chronic maintenance or suppressive therapy
* HIV negative

Other

* No retinitis or choroiditis
* No history of seizures
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy (e.g., interleukins, interferons, melanoma vaccines, IV immunoglobulin, or expanded polyclonal tumor-infiltrating lymphocytes or lymphokine-activated killer therapy)

Chemotherapy

* At least 4 weeks since prior chemotherapy (standard or experimental) and recovered

Endocrine therapy

* No concurrent systemic steroids except for toxicity management

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* At least 4 weeks since prior immunosuppressive therapy
* More than 4 weeks since prior experimental drugs and recovered
* No concurrent pentoxifylline
* No other concurrent investigational agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2001-11; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassian Yee, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States